CLINICAL TRIAL: NCT01331941
Title: An Open-label Pharmacokinetic Study of AMG 386 in Advanced Cancer Subjects With Normal and Impaired Renal Function
Brief Title: A Pharmacokinetic Study of AMG 386 in Cancer Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090277
Record Dates: First submitted 2011-03-24; First posted 2011-04-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Advanced Solid Tumors; Kidney Disease; Renal Impairment
Keywords: AMG 386; Pharmacokinetic; Renal Impairment
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — trebananib; Paclitaxel

ARMS (4):
- Group 1 (Experimental): Cancer subjects with normal renal function.
  Interventions: Drug: AMG 386 + Paclitaxel; Drug: AMG 386
- Group 3 (Experimental): Cancer subjects with moderate renal impairment.
  Interventions: Drug: AMG 386 + Paclitaxel; Drug: AMG 386
- Group 4 (Experimental): Cancer subjects with severe renal impairment.
  Interventions: Drug: AMG 386
- Group 2 (Experimental): Cancer subjects with mild renal impairment.
  Interventions: Drug: AMG 386 + Paclitaxel; Drug: AMG 386

INTERVENTIONS:
Drug: AMG 386 + Paclitaxel — 15 mg/kg IV (in the vein) of AMG 386 weekly + 80 mg/m^2 IV (in the vein) 3 weeks on/1 week off, optional beginning week 6 until progression, unacceptable toxicity, or withdrawal of consent.
  Arms: Group 1; Group 2; Group 3
Drug: AMG 386 — 15 mg/kg IV (in the vein) weekly beginning week 1 day 1 until progression, unacceptable toxicity, or withdrawal of consent.

SUMMARY:
This is a phase 1, open-label pharmacokinetic study where up to 40 subjects with advanced solid tumors (up to 6-10 with normal renal function and up to 18-30 with varying degrees of renal dysfunction) will receive weekly doses of AMG 386 intravenously. The primary objective is to evaluate the pharmacokinetics (PK) of single agent AMG 386 in subjects with various degrees of renal function. Once the AMG 386 PK characterization is complete in the first 5 weeks of the study, all subjects will be allowed to continue to receive AMG 386 weekly only or subjects in group 1, 2 or 3 can opt to receive AMG 386 weekly in combination with paclitaxel until disease progression, unacceptable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age
* Must have a pathologically documented, and definitively diagnosed, advanced solid tumor that is refractory to standard treatment, or for which no curative therapy is available, or for subjects who refuse standard therapy
* Evaluable OR measurable disease by RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Life expectancy of > 3 months, in the opinion of and as documented by the investigator
* Subject or subject's legally acceptable representative has provided informed consent

Exclusion Criteria:

* Subjects with gastric cancer or any malignancy with purely squamous cell histology
* Known history of primary central nervous system (CNS) tumors or CNS metastases
* Myocardial infarction within 1 year before study day 1, unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association > class II, uncontrolled hypertension [diastolic > 90 mmHg; systolic > 150 mmHg in repeated measurements])
* History of stroke, arterial or venous thrombosis, or pulmonary embolism within 1 year before study day 1
* Active grade 2 or greater peripheral vascular disease or peripheral edema
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis)
* Non-healing wound, ulcer (including gastrointestinal) or fracture
* Known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection
* Major surgery within 4 weeks before study day 1
* Absolute neutrophils count (ANC) < 1.0 x 10^9/L; or platelet count < 100 x 10^9/L; or hemoglobin < 9 g/dL; or PTT / aPTT > 1.5 x institutional upper limit of normal (ULN) ); or INR > 1.5
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN (> 5.0 x ULN if liver metastases present)
* Alkaline phosphatase > 2.5 x ULN (> 5.0 x ULN if attributable to liver or bone metastasis)
* Total bilirubin > 1.5 x ULN
* Other investigational procedures during the study
* Previous anti-cancer therapy or investigational agent within 4 weeks prior to study day 1
* Anticoagulation therapy within 4 weeks of study day 1 and while on study (except low dose warfarin (≤ 2 mg/kg) for prophylaxis against central venous catheter thrombosis)
* Men and women of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study and an additional 6 months after the last dose of AMG 386. Highly effective methods of birth control include sexual abstinence (men, women); vasectomy or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or IUD (women).
* Women who are lactating/breastfeeding.
* Women with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2013-02-26 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve (AUC) | Week 1-5.
Maximum observed concentration (Cmax) | Week 1-5.
Time to maximum concentration (tmax) | Week 1-5.
Minimum observed concentration (Cmin) | Week 1-5.
Clearance (CL) of AMG 386 calculated as dose divided by AUC on week 5. | Week 1-5

SECONDARY OUTCOMES:
Adverse events as a measure of safety | Weekly at each visit AMG 386 is administered, on day 30, 31 and 32 when only PK assessments are scheduled up to and including the last study visit 30 days after the last AMG 386 administration.
Changes in vital signs as a measure of safety | Weekly at each visit AMG 386 is administered up to and including the last study visit 30 days after the last AMG 386 administration.
Changes in clinical laboratory tests as a measure of safety | Weekly from week 1-9 then every 4 weeks thereafter including the last study visit 30 days after the last AMG 386 administration.
Anti-AMG 386 antibody formation | Week 1, week 5, week 9 and every 16 weeks thereafter including the last study visit 30 days after the last AMG 386 administration.
Tumor objective response measured by CT or MRI (without Gadolinium contrast agents) and assessed by RECIST 1.1 criteria. | Week 5 and every 8 weeks thereafter until the subject's end of participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lebanon, New Hampshire
  - Research Site, Cleveland, Ohio

REFERENCES:
- [Background] Wu B, Lewis LD, Harvey RD, Rasmussen E, Gamelin E, Sun YN, Friberg G, Koyner JL, Dowlati A, Maitland ML. A Pharmacokinetic and Safety Study of Trebananib, an Fc-Fusion Peptibody, in Patients With Advanced Solid Tumors and Varying Degrees of Renal Dysfunction. Clin Pharmacol Ther. 2017 Aug;102(2):313-320. doi: 10.1002/cpt.617. Epub 2017 Jun 9. PMID 28074547
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com